CLINICAL TRIAL: NCT00054275
Title: A Phase II Study Of The Weekly Administration Of Docetaxel In Combination With The Epidermal Growth Factor Receptor Inhibitor OSI-774 In Recurrent And/Or Metastatic Breast Cancer
Brief Title: Erlotinib Plus Docetaxel in Treating Patients With Stage IV or Recurrent Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paula Silverman, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Paula Silverman, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1102; P30CA043703 (NIH); 07-02-14M (Other: University Hospitals IRB); CASE-CWRU-1102 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Docetaxel; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib Plus Docetaxel (Experimental)
  Interventions: Drug: docetaxel; Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: docetaxel — Docetaxel IV infusion weekly for 3 weeks with a one-week break. One cycle is 4 weeks (28 days). Patients' actual weight will be used to calculate dose.
  Other Names: Taxotere; RP 56976; NSC #628503
Drug: erlotinib hydrochloride — OSI-774 will be taken 1 hour before or 2 hours after meals. Cycle 1 will be administered at dose level -1.If no grade 3 or 4 toxicity occurs during cycle 1, then the patient may proceed to be treated at dose level 0 for the remaining chemotherapy cycles.
  Other Names: CP-358; 774; USAN: erlotinib hydrochloride; Tarceva

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining erlotinib with docetaxel may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining erlotinib with docetaxel in treating patients who have stage IV or recurrent breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor effects of erlotinib and docetaxel, in terms of objective response, stabilization of disease, and progression-free survival, in patients with stage IV or recurrent breast cancer.
* Determine time to tumor progression in patients treated with this regimen.
* Compare time to tumor progression in patients who achieve disease stabilization or response after treatment with this regimen and continue to receive erlotinib versus patients who do not receive additional erlotinib.

OUTLINE: Patients receive docetaxel IV over 1 hour once weekly for 3 weeks and oral erlotinib once daily beginning on day 1. Treatment repeats every 4 weeks for a minimum of 6 courses in the absence of unacceptable toxicity or disease progression. Patients achieving maximal tumor response or stabilization of disease after 6 courses may continue to receive erlotinib alone until disease progression.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 12-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV or recurrent adenocarcinoma of the breast
* Measurable disease
* Disease recurrence must not be within 1 year of receiving prior adjuvant docetaxel
* Stable brain metastases allowed
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Male or female

Menopausal status

* Not specified

Performance status

* ECOG (Eastern Cooperative Oncology Group) 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 6 months

Hematopoietic

* WBC(White Blood Count) at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin at least 8 g/dL

Hepatic

* Bilirubin normal
* AST(aspartate aminotransferase)/ALT(alanine aminotransferase) no greater than 2.5 times upper limit of normal

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min
* No clinically significant proteinuria
* No significant impairment of renal function

Cardiovascular

* No New York Heart Association class III or IV heart disease
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No inadequately controlled hypertension

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No prior severe hypersensitivity reaction to docetaxel or drugs formulated with polysorbate 80
* No other malignancy within the past 10 years except inactive nonmelanoma skin cancer, carcinoma in situ of the cervix, carcinoma in situ of the breast, or bilateral breast cancer
* No ongoing or active infection
* No peripheral neuropathy greater than grade 1
* No other concurrent uncontrolled medical condition that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior trastuzumab (Herceptin) allowed

Chemotherapy

* See Disease Characteristics
* No prior chemotherapy for recurrent or metastatic disease
* Prior adjuvant chemotherapy allowed

Endocrine therapy

* Prior hormonal therapy allowed

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2002-12; Primary Completion 2010-04 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Silverman, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from University Hospitals and its satellite hospitals from 12/4/2002 through 9/22/2006.
Groups:
- Docetaxel and OSI-774: docetaxel IV over 1 hour once weekly for 3 weeks and oral erlotinib once daily
Period: Overall Study
Arm/Group | Docetaxel and OSI-774
Started | 39
Completed | 28
Not Completed | 11
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 5
Not completed — Progressive disease in cycle 1 | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel and OSI-774
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 51 [28 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Disease Response (Tumor Measurements)Per RECIST Criteria v. 2000
Description: Response and progression will be evaluated in this study using the criteria by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria. Partial Response: At least a 30% decrease in the sum of the longest diameter (LD) of target lesions. Progressive Disease: At least a 20% increase in the sum of the LD of target lesions. Stable Disease: Neither sufficient shrinkage nor sufficient increase.
Time Frame: after 6 course (6 months) of combination therapy
Population: Excluding 11 not evaluable cases
Measure: Number; unit: participants
Arm/Group | Docetaxel and OSI-774
Number analyzed (Participants) | 28
participants
  Partial response | 11 [0.23 to 0.58]
  Disease progression | 14
  Stable disease | 3
Statistical Analysis 1: Comparison: Docetaxel and OSI-774; Test type: Superiority or Other; p = 0.95, confidence interval for partial response; Confidence interval for partial response rate using Wilson's Method; proportion of pts with partial response = 0.39, 95% CI 2-sided [0.23 to 0.58]

2. Secondary Outcome: Progression Free Survival(PFS)
Description: Progression free survival was defined as time from the start of treatment to the date of cancer progression, or death, and censored at the date of last follow-up for those without disease progression and still alive. Stable disease is measured from the start of the treatment until progression, taking as reference the smallest measurements recorded since the treatment started. Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel and OSI-774
Number analyzed (Participants) | 39
months | 8.4 [4.8 to 12.8]

3. Secondary Outcome: Overall Survival as of 2008
Description: Overall survival (OS) was defined as time from the start of treatment to death, and censored at the time of last assessment for survivors.
Time Frame: 5 yrs
Population: Including 10 patients with only 1 cycle of treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel and OSI-774
Number analyzed (Participants) | 39
months | 22.3 [15.2 to 30.6]

ADVERSE EVENTS:
Time Frame: Patients will be evaluated for adverse events at each study visit for the duration of their participation in the study and for 30 days after the discontinuation of Tarceva.
Arm/Group | Docetaxel and OSI-774
Serious Adverse Events (participants affected / at risk) | 28/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel and OSI-774 (N=39)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 5
Bone Pain (Musculoskeletal and connective tissue disorders) | 2
Cerebrovascular Ischemia (Nervous system disorders) | 1
Chest Pain (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Eye tearing (Eye disorders) | 1
Fatigue (General disorders) | 6
Headache (Nervous system disorders) | 1
Hyperbilirubinbemia (Investigations) | 1
Hyperbilirubinemia (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infection (Infections and infestations) | 2
Leukopenia (Blood and lymphatic system disorders) | 4
Light headedness (Nervous system disorders) | 1
Lymphopenia (Investigations) | 14
Mucositis (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 4
Pericarditis (Cardiac disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
SGOT (AST) (Investigations) | 1 — serum glutamic-oxaloacetic transaminase
SGPT (ALT) (Investigations) | 2 — serum glutamic-pyruvic transaminase
Sinus Tach. (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Taste Change(dysgeusia) (Nervous system disorders) | 1
Vaginitis (Reproductive system and breast disorders) | 1
Vomiting (Gastrointestinal disorders) | 1 — Emesis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel and OSI-774 (N=39)
Abdominal Pain (Gastrointestinal disorders) | 2
Alkaline Phosphatase (Investigations) | 14
Alopecia (Skin and subcutaneous tissue disorders) | 24
Anemia (Blood and lymphatic system disorders) | 28
Anorexia (Metabolism and nutrition disorders) | 28
Anxiety (Psychiatric disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bicarbonate (Metabolism and nutrition disorders) | 9
Bilirubin (Investigations) | 4
Blurred Vision (Eye disorders) | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 7
Bruising (Injury, poisoning and procedural complications) | 3
Conjunctivitis (Eye disorders) | 5
Constipation (Gastrointestinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 3
Depression (Psychiatric disorders) | 4
Derm (Skin and subcutaneous tissue disorders) | 3
Diarrhea (Gastrointestinal disorders) | 27
Dizziness (Nervous system disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 10
Dry eye (Eye disorders) | 3
Dysgeusia (Nervous system disorders) | 18 — Taste change
Dysphagia (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12
Dysuria (Renal and urinary disorders) | 3 — Painful urination
Edema (General disorders) | 6
Emesis (Gastrointestinal disorders) | 9 — vomiting
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 — Bleeding from the nose
Fatigue (General disorders) | 37
Fever (General disorders) | 4
Flushing (Vascular disorders) | 4
Frequent urination (Renal and urinary disorders) | 3
Hand-Foot syndrome (Skin and subcutaneous tissue disorders) | 4
Headache (Nervous system disorders) | 5
Hot Flashes (Vascular disorders) | 17
Hyperbilirubinemia (Investigations) | 10
Hyperglycemia (Metabolism and nutrition disorders) | 13
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 17
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 10
Hypokalemia (Metabolism and nutrition disorders) | 15
Hypomagnesmia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 10
Infection (General disorders) | 8
Injection site reaction (General disorders) | 2
Insomnia (Psychiatric disorders) | 15
Leg edema (General disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 23
Light headedness (Nervous system disorders) | 10
Lymphedema (Vascular disorders) | 2
Lymphopenia (Investigations) | 24
Mucositis (Gastrointestinal disorders) | 22
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 10
Nail Changes (Skin and subcutaneous tissue disorders) | 10
Nausea (Gastrointestinal disorders) | 27
Neuropathy (Nervous system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 15
Odynophagia (Gastrointestinal disorders) | 4 — Painful swallowing
Pain (General disorders) | 11
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5
Pruritis (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 27
Reflux (Gastrointestinal disorders) | 7
Rigors or chills (General disorders) | 4
SGOT (AST) (Investigations) | 18
SGPT (ALT) (Investigations) | 17
Sensory Neuropathy (Nervous system disorders) | 13
Stomatitis (Gastrointestinal disorders) | 4
Stridor (Respiratory, thoracic and mediastinal disorders) | 4
Tearing (Eye disorders) | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Vaginitis (Reproductive system and breast disorders) | 2
Weight Loss (Investigations) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes